CLINICAL TRIAL: NCT02411318
Title: Influence of Lifestyle Factors on Neutrophil Migration Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-0218; A194200 (Other: UW Madison); ENGR\BIOMEDICAL ENGR (Other: UW Madison)
Record Dates: First submitted 2015-03-25; First posted 2015-04-08 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-03

CONDITIONS: Neutrophil Chemotactic Response
MeSH Terms: interventions — Exercise; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cardiovascular Exercise (Experimental): Participants will ride a stationary bike and maintain their target heart rate (according to the American Heart Association guidelines) for 30 minutes. For example, a 30 year old will have a target heart rate zone of 95-162 beats per minute. A baseline blood sample will be acquired before the participant begins exercising. In the following 30 minutes, participants will ride the exercise bike, and their heart rate and general status will be assessed continuously. Specifically, heart rate will be monitored using a chest strap heart rate monitor. Two additional lancet punctures will be performed after the exercise to measure the changes in neutrophil function: one immediately following the 30 minute exercise period and one 30 minutes after the exercise has been completed.
  Interventions: Behavioral: Exercise
- Caffeine Consumption (Experimental): Participants will be exposed to a moderate dose of caffeine (200 mg capsule in one sitting) from a common commercial product. After consent and screening, a baseline blood sample will be acquired using the lancet puncture procedure. The participant will then be instructed to swallow a 200 mg caffeine capsule. Two additional lancet punctures will be performed after the caffeine ingestion: one after 30 minutes post-ingestion and another one after 60 minutes.
  Interventions: Drug: ProLab 200mg caffeine capsule
- Ethanol Ingestion (Experimental): Participants will be weighed and their required alcohol dose determined according to the equation used by the Madison Police Department during alcohol training workshops: 1 mL of 80 proof (40%) alcohol per pound of body weight. Participants will be permitted to consume the drink at their own pace, although no slower than one drink per hour. Breath Alcohol Concentration (BAC) will be tested 20 minutes after drinking has ceased in order to clear mouth alcohol that may affect the BAC reading. Participants at 0.05 BAC and above will have blood drawn via lancet puncture. In addition to the lancet puncture done once the alcohol level is reached, an additional lancet puncture will be performed 1 hour later.
  Interventions: Other: Ethanol ingestion
- Glucose Ingestion (Experimental): After a baseline blood sample is acquired, participants will consume 100 grams of glucose within 5 minutes. Two additional lancet punctures will be performed after the glucose ingestion, one at 30 minutes post-ingestion, and one at 60 minutes post-ingestion.
  Interventions: Drug: Glucose Tolerance Drink
- Glucose and Caffeine Ingestion (Experimental): After a baseline blood sample is acquired, participants will swallow 200mg of caffeine in capsule form and consume 100 grams of glucose within 5 minutes. Two additional lancet punctures will be performed after the caffeine and glucose ingestion, one at 30 minutes post-ingestion, and one at 60 minutes post-ingestion.
  Interventions: Drug: ProLab 200mg caffeine capsule; Drug: Glucose Tolerance Drink

INTERVENTIONS:
Behavioral: Exercise — Participants will ride a stationary bike and maintain their target heart rate (according to the American Heart Association guidelines) for 30 minutes.
  Arms: Cardiovascular Exercise
Drug: ProLab 200mg caffeine capsule — Participants will swallow one ProLab caffeine 200mg tablet.
  Arms: Caffeine Consumption; Glucose and Caffeine Ingestion
Other: Ethanol ingestion — Participants will consume a dose of 80 proof alcohol according to their body weight to reach a breath alcohol concentration of 0.05.
  Arms: Ethanol Ingestion
Drug: Glucose Tolerance Drink — Participants will consume 100 grams of glucose
  Arms: Glucose Ingestion; Glucose and Caffeine Ingestion

SUMMARY:
This study will determine how common lifestyle practices affect the behavior of neutrophils (a type of immune cell) at shorter time scales than previously possible.

DETAILED DESCRIPTION:
This study will investigate how external factors implicated in immunity such as exercise, caffeine ingestion, ethanol, glucose, and glucose and caffeine ingestion influence neutrophil migration.

Neutrophils are the most prominent immune cell in human blood and are involved in a complex equilibrium of immune protection and autoimmune damage. Their recruitment to an inflammatory or wounding site is controlled by the sensing and directed migration to a concentration gradient of attractant molecules, a process called chemotaxis. Immune cells are also implicated in many diseases including cancer. The ability to measure the amplitude of a response over time for a specific patient, and the variation of this response when the patient engages in certain activities or consumes certain substances will improve understanding of how certain lifestyle factors impact the immune response. Traditional assays require large volumes of blood and a long purification process, which may affect neutrophil function and strictly limits the number of draws possible from a single patient. The novel microfluidic assay proposed limits these drawbacks as it has the capability to purify neutrophils from a 3 µL drop of blood in less than 5 minutes and measure their chemotaxis in a gradient of chemokines. Critically, the proposed studies will begin to fill a gap in current understanding of immune response as previous studies focused on single endpoints likely missing early events in the response to external stimulus. Understanding this temporal response may have implications in the development of new treatments as well as improvements in diagnosis of improper immune response.

The KOALA (Kit On A Lid Assay) approach was developed in Professor Dave Beebe's lab and has been validated in a mouse model and in human asthmatic patients. In a collaboration with Dr. Anna Huttenlocher, it has been shown that, in contrast to traditional neutrophil purification, KOALA can be performed with small volumes of blood, and a much quicker purification time.

Due to its unique qualities, KOALA allows for repeated evaluation of neutrophil adhesion and chemotaxis properties, thus making it an attractive method for studying dynamic neutrophil changes that may occur as a result of an external factor.

Using traditional macrobiology tools, researchers have identified several factors that may play important roles in reducing neutrophil responsiveness and migration ability. Lifestyle and diet factors, amongst others, have been shown to impact neutrophil count, migration and biochemical function. For example, sleep deprivation has been linked with higher neutrophil count, despite a known immuno-depressive effect. Physical exercise results in increased neutrophil counts and increased neutrophil degranulation. Dietary factors, such as caffeine and ethanol have been shown to impact immune function.

Blood glucose will be tested at each time point using a blood glucose monitor to determine whether the lifestyle factor is affecting blood glucose (and consequently, neutrophil function). Alcohol consumption can cause both high and low blood sugar. Specifically, while low doses of alcohol may have a protective effect against risk of diabetes and metabolic syndrome, heavy drinking has been associated with higher glucose levels, resulting in increased risk of both diabetes and metabolic syndrome. Similarly, acute ingestion of caffeine has been shown to increase blood glucose levels, but several epidemiological studies have shown regular coffee consumption in associated with a lower risk of type 2 diabetes. Measuring blood glucose on subjects in the glucose study may show dose dependent effects on neutrophils.

To build on this research, the investigators intend to probe the role of these lifestyle factors on neutrophil migration over much shorter time scales than has been previously studied. The investigators propose to examine the effects of exercise, ethanol ingestion and caffeine consumption on neutrophil behavior.

Whole blood obtained from subjects by finger stick will be used in KOALA to isolate neutrophils. Neutrophil function will be assessed by measuring absolute migration speed, chemotactic index and chemotaxis velocity (directional velocity toward the formation of the gradient of chemoattractant).

The primary outcome of this study will be to determine whether exercise, caffeine consumption, ethanol, glucose and combined glucose and caffeine ingestion affect neutrophil chemotactic velocity. The secondary outcomes are to determine whether exercise, caffeine consumption, ethanol, glucose and combined glucose and caffeine ingestion affect the absolute speed and chemotactic index of neutrophils. The investigators will also assess whether cytokine profiles in the blood change as a result of engaging int he specified lifestyle factors.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent and ability to speak and read English.
* Male or female with no chronic or acute health concerns that might affect subject safety during the study or interfere with the study results
* No intake of medication that the researchers believe will significantly influence immune function in the 48 hours proceeding the lancet puncture (examples given in the section entitled "Exclusion Criteria")
* In good physical health
* Regularly exercise at least 30 minutes 3 times per week (exercise cohort)

Exclusion Criteria:

* Currently participating in another clinical trial
* History of significant systemic disease (eg. cancer, infection, hematological, renal, hepatic, coronary artery disease or other cardiovascular disease, endocrinologic, neurologic, rheumatologic, or gastrointestinal disease)
* Use of beta blockers or corticosteroids
* Currently taking medications that are not recommended to be taken in conjunction with alcohol
* Acute illness or evidence of clinically significant active infection
* Currently receiving immunotherapy
* Pregnant women
* Ingested medication (e.g. systemic corticosteroids) within 48 hours preceding the draw that the researchers believe may have an effect on immune response or the immune system
* Performed any activity that conflicts (eg. drinking any alcohol prior to the study), in the judgment of the investigator, with the external factor to be tested in the study (if any)
* Alcoholic or other health conditions for which alcohol consumption is contraindicated
* Consume more than 7 drinks per week (women alcohol cohort)
* Consume more than 14 drinks per week (men alcohol cohort)
* Consume more than three (8 oz.) servings of coffee, caffeinated soft drinks/tea (12 oz.) per day (caffeine cohort)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2014-09-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Exercise-Related Neutrophil Chemotactic Velocity | baseline, 30 min, 60 min
  Participants will ride a stationary bike and maintain their target heart rate for 30 min. Blood samples via lancet will be collected at baseline, 30 min (immediately post intervention), and 60 min.
Change in Caffeine-Related Neutrophil Chemotactic Velocity | baseline, 30 min, 60 min
  Participants will consume a moderate dose of caffeine via 200mg capsule. Blood samples via lancet will be collected at baseline, 30 min (immediately post intervention), and 60 min.
Change in Ethanol-Related Neutrophil Chemotactic Velocity | baseline, 1-3 hours from baseline, up to 2-4 hours from baseline
  Participants will consume a weight-calculated dose of alcohol sufficient to increase their blood alcohol concentration (BAC) to 0.05. Blood samples via lancet will be collected at baseline, 1-3 hours (when BAC reached 0.05) and 1 hour after previous collection.
Change in Glucose-Related Neutrophil Chemotactic Velocity | baseline, 30 min, 60 min
  Participants will consume 100g glucose tolerance drink within 5 minutes. Blood samples via lancet will be collected at baseline, 30 min (immediately post intervention), and 60 min.
Change in Caffeine Plus Glucose-Related Neutrophil Chemotactic Velocity | baseline, 30 min, 60 min
  Participants will consume a moderate dose of caffeine via 200mg capsule and 100g of glucose tolerance drink within 5 min. Blood samples via lancet will be collected at baseline, 30 min (immediately post intervention), and 60 min.

SECONDARY OUTCOMES:
Change in Exercise-Related Neutrophil Absolute Speed | baseline, 30 min, 60 min
  Participants will ride a stationary bike and maintain their target heart rate for 30 min. Blood samples via lancet will be collected at baseline, 30 min (immediately post intervention), and 60 min.
Change in Exercise-Related Neutrophil Chemotactic Index | baseline, 30 min, 60 min
  Participants will ride a stationary bike and maintain their target heart rate for 30 min. Blood samples via lancet will be collected at baseline, 30 min (immediately post intervention), and 60 min.
Change in Caffeine-Related Neutrophil Absolute Speed | baseline, 30 min, 60 min
  Participants will consume a moderate dose of caffeine via 200mg capsule. Blood samples via lancet will be collected at baseline, 30 min (immediately post intervention), and 60 min.
Change in Caffeine-Related Neutrophil Chemotactic Index | baseline, 30 min, 60 min
  Participants will consume a moderate dose of caffeine via 200mg capsule. Blood samples via lancet will be collected at baseline, 30 min (immediately post intervention), and 60 min.
Change in Ethanol-Related Neutrophil Absolute Speed | baseline, 1-3 hours from baseline, up to 2-4 hours from baseline
  Participants will consume a weight-calculated dose of alcohol sufficient to increase their blood alcohol concentration (BAC) to 0.05. Blood samples via lancet will be collected at baseline, 1-3 hours (when BAC reached 0.05) and 1 hour after previous collection.
Change in Ethanol-Related Neutrophil Chemotactic Index | baseline, 1-3 hours from baseline, up to 2-4 hours from baseline
  Participants will consume a weight-calculated dose of alcohol sufficient to increase their blood alcohol concentration (BAC) to 0.05. Blood samples via lancet will be collected at baseline, 1-3 hours (when BAC reached 0.05) and 1 hour after previous collection.
Change in Glucose-Related Neutrophil Absolute Speed | baseline, 30 min, 60 min
  Participants will consume 100g glucose tolerance drink within 5 minutes. Blood samples via lancet will be collected at baseline, 30 min (immediately post intervention), and 60 min.
Change in Glucose-Related Neutrophil Chemotactic Index | baseline, 30 min, 60 min
  Participants will consume 100g glucose tolerance drink within 5 minutes. Blood samples via lancet will be collected at baseline, 30 min (immediately post intervention), and 60 min.
Change in Caffeine Plus Glucose-Related Neutrophil Absolute Speed | baseline, 30 min, 60 min
  Participants will consume a moderate dose of caffeine via 200mg capsule and 100g of glucose tolerance drink within 5 min. Blood samples via lancet will be collected at baseline, 30 min (immediately post intervention), and 60 min.
Change in Caffeine Plus Glucose-Related Neutrophil Chemotactic Index | baseline, 30 min, 60 min
  Participants will consume a moderate dose of caffeine via 200mg capsule and 100g of glucose tolerance drink within 5 min. Blood samples via lancet will be collected at baseline, 30 min (immediately post intervention), and 60 min.

CONTACTS AND LOCATIONS:
Overall Officials: David J Beebe, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Background] Bagby GJ, Zhang P, Stoltz DA, Nelson S. Suppression of the granulocyte colony-stimulating factor response to Escherichia coli challenge by alcohol intoxication. Alcohol Clin Exp Res. 1998 Nov;22(8):1740-5. PMID 9835289
- [Background] Bird MD, Zahs A, Deburghgraeve C, Ramirez L, Choudhry MA, Kovacs EJ. Decreased pulmonary inflammation following ethanol and burn injury in mice deficient in TLR4 but not TLR2 signaling. Alcohol Clin Exp Res. 2010 Oct;34(10):1733-41. doi: 10.1111/j.1530-0277.2010.01260.x. Epub 2010 Jul 1. PMID 20608903
- [Background] Boe DM, Nelson S, Zhang P, Quinton L, Bagby GJ. Alcohol-induced suppression of lung chemokine production and the host defense response to Streptococcus pneumoniae. Alcohol Clin Exp Res. 2003 Nov;27(11):1838-45. doi: 10.1097/01.ALC.0000095634.82310.53. PMID 14634502
- [Background] Boudjeltia KZ, Faraut B, Stenuit P, Esposito MJ, Dyzma M, Brohee D, Ducobu J, Vanhaeverbeek M, Kerkhofs M. Sleep restriction increases white blood cells, mainly neutrophil count, in young healthy men: a pilot study. Vasc Health Risk Manag. 2008;4(6):1467-70. doi: 10.2147/vhrm.s3934. PMID 19337560
- [Background] Chimenti L, Morici G, Paterno A, Santagata R, Bonanno A, Profita M, Riccobono L, Bellia V, Bonsignore MR. Bronchial epithelial damage after a half-marathon in nonasthmatic amateur runners. Am J Physiol Lung Cell Mol Physiol. 2010 Jun;298(6):L857-62. doi: 10.1152/ajplung.00053.2010. Epub 2010 Apr 2. PMID 20363849
- [Background] Horrigan LA, Kelly JP, Connor TJ. Caffeine suppresses TNF-alpha production via activation of the cyclic AMP/protein kinase A pathway. Int Immunopharmacol. 2004 Oct;4(10-11):1409-17. doi: 10.1016/j.intimp.2004.06.005. PMID 15313438
- [Background] Sackmann EK, Berthier E, Young EW, Shelef MA, Wernimont SA, Huttenlocher A, Beebe DJ. Microfluidic kit-on-a-lid: a versatile platform for neutrophil chemotaxis assays. Blood. 2012 Oct 4;120(14):e45-53. doi: 10.1182/blood-2012-03-416453. Epub 2012 Aug 22. PMID 22915642
- [Background] Sackmann EK, Berthier E, Schwantes EA, Fichtinger PS, Evans MD, Dziadzio LL, Huttenlocher A, Mathur SK, Beebe DJ. Characterizing asthma from a drop of blood using neutrophil chemotaxis. Proc Natl Acad Sci U S A. 2014 Apr 22;111(16):5813-8. doi: 10.1073/pnas.1324043111. Epub 2014 Apr 7. PMID 24711384